CLINICAL TRIAL: NCT05630469
Title: Prediction of Antidepressant Effects of Electroconvulsive Therapy
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Pia Baldinger-Melich, Assoc.Prof., Medical University of Vienna
Other Study IDs: KLI 1098-B
Record Dates: First submitted 2022-11-10; First posted 2022-11-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Depressive Disorder, Major
Keywords: electroconvulsive therapy; neuroimaging; response prediction; biomarker
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Depression: Depressive patients (pharmaco-resistant) undergoing electroconvulsive therapy
  Interventions: Other: Electroconvulsive therapy

INTERVENTIONS:
Other: Electroconvulsive therapy — repetitive induction of a generalized seizure under controlled conditions (muscle relaxation and sedation)

SUMMARY:
Despite its successful use for more than 80 years, the mechanisms of action of electroconvulsive therapy (ECT) are still not fully understood. ECT has been shown to be accompanied by changes in regional brain volumes and connectivity measures, as well as biochemical alterations. However, how these changes relate to ECT response remains to be further elucidated; up to now, there are no objective markers for the targeted use of ECT in clinical practice.

Methods: Study design: longitudinal mono-centre study with duration of 36 months. Subjects: 30 depressed patients (aged 18-65 years) eligible for ECT. Measurements: subjects will undergo 2 3-Tesla MRI scans (one before and one after a course of ECT), including structural MRI, resting-state functional MRI, task-based functional MRI and MR spectroscopy. Blood, CSF sampling and clinical assessments will be performed once before and once after the ECT course. ECT: Each patient will be treated in a min. of 8 bitemporal ECT sessions (~4 weeks). Data analysis: Longitudinal changes in brain imaging parameters and laboratory measures (before/after ECT) will be assessed using repeated-measures analysis of covariance. Machine learning with random forests will be employed to identify a pattern of pretreatment imaging, biochemical (serum and CSF) and clinical parameters that are best qualified to predict response to ECT as defined by a reduction of ≥50% of baseline HAMD17.

Hypotheses: 1. ECT will be accompanied by changes in brain morphology, functional connectivity, neuronal activation in response to cognitive and reward-related stimuli and neurochemical signals in the brain. 2. ECT leads to changes in blood- and CSF-based markers of neuronal plasticity, neurodegeneration and inflammation, as well as genetic/epigenetic markers. 3. Predictive markers of ECT response can be established based on the relationships between imaging, neurochemical and clinical markers and treatment response.

Innovation: This study would be the first to combine multimodal MRI measures with the assessment of biomarkers in the CSF in the context of ECT. The implementation of the proposed trial represents an important step towards a better understanding of the powerful antidepressant properties of ECT. By relating treatment effects and potentially underlying biological mechanisms on numerous complementary levels, the study might help to identify biomarkers that distinguish patients who are likely to benefit from ECT from non-responders. Ultimately, results of the study might be useful in order to establish an individualized medical indication for ECT.

ELIGIBILITY:
Inclusion Criteria:

* male or female inpatients (18-65 years old)
* ICD-10 diagnosis of severe unipolar depression (F32.2, F32.3, F33.2, F33.3)
* HAMD17 ≥ 23
* physical health
* ability to understand and willingness to sign the written informed consent document
* negative drug screening, negative urine pregnancy test in women
* antidepressant and antipsychotic medication in steady state for at least 10 days prior inclusion
* anesthesiological approval for ECT

Excusion criteria:

* severe somatic or neurological disease
* current comorbid psychiatric disorder, including bipolar depression (according to DSM-5)
* current or past history of schizophrenia or schizoaffective disorder
* current use of alcohol, drugs of abuse, or any medication in a manner which is indicative of chronic abuse or who meet DSM-5 criteria for alcohol or other substance dependence
* clinically relevant abnormalities on a general physical examination and routine laboratory screening
* pregnancy, breast feeding
* contraindications to lumbar puncture (increased intracranial volume, anticoagulant medication, uncorrected bleeding diathesis, coagulopathy, congenital spine abnormality, recent spinal trauma/surgery, skin infection at puncture site)
* any implant or stainless steel graft contraindicated for MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with a major depressive episode (unipolar depression) as determined by a structured clinical interview for DSM-5 (SCID-5-clinical version) and the 17-item Hamilton rating scale for depression (HAM-D score ≥ 23) who did not respond to conventional pharmacological antidepressant treatment and are eligible for ECT will be recruited at the Department of Psychiatry and Psychotherapy at the General Hospital of Vienna.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
imaging parameter - sMRI | 3 years
  cortical thickness
imaging parameters - DTI | 3 years
  mean diffusivity
imaging parameters - fMRI | 3 years
  BOLD activity (task-based fMRI for cognition and anhedonia)
imaging parameters - rsfMRI | 3 years
  BOLD activity (rsfMRI)
imaging parameters - MRS | 3 years
  Glx, NAA and GABA concentrations (MRS)
biochemical parameters - neurodegeneration | 3 years
  concentrations of markers of neurodegeneration serum and CSF
biochemical parameters - inflammation | 3 years
  concentrations of markers of neuroinflammation serum and CSF
biochemical parameters - neurplasticity | 3 years
  concentrations of markers of neuroplasticity serum and CSF
response prediction | 3 years
  machine learning - how do outcome 1 and 2 relate to response to ECT

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided